CLINICAL TRIAL: NCT06353555
Title: A Study on the Efficacy of Thyroid Hormone Replacement Therapy for Secondary Hypothyroidism Following Intracerebral Hemorrhage
Brief Title: Efficacy of Thyroid Hormone Replacement for Secondary Hypothyroidism Following Intracerebral Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wei Junji, clinical professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUMCH-20240311
Record Dates: First submitted 2024-03-11; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Intracerebral Hemorrhage; Low T3 Syndrome; Neurocritical Care; Hormone Replacement Therapy
MeSH Terms: conditions — Cerebral Hemorrhage; Euthyroid Sick Syndromes | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyroid hormone replacement therapy (Experimental): Upon discovering low T3 or low T4 levels, administer oral levothyroxine sodium tablets daily. If accompanied by a decrease in TSH, the regimen is 100μg qd (for individuals weighing <75kg) or 150μg qd (for individuals weighing >75kg). If not accompanied by a decrease in TSH, the regimen is 50μg qd. However, if thyroid function does not significantly improve within 3 days of medication, the regimen is adjusted to 100μg qd. Treatment should continue until transfer out of the NICU or discharge, with a minimum duration of 7 days.
  Interventions: Drug: Euthyrox
- Non-thyroid hormone replacement therapy (Sham Comparator): Patients will not receive the oral levothyroxine sodium tablets.
  Interventions: Drug: Euthyrox

INTERVENTIONS:
Drug: Euthyrox — Upon discovering low T3 or low T4 levels, administer oral levothyroxine sodium tablets daily. If accompanied by a decrease in TSH, the regimen is 100μg qd (for individuals weighing <75kg) or 150μg qd (for individuals weighing >75kg). If not accompanied by a decrease in TSH, the regimen is 50μg qd. However, if thyroid function does not significantly improve within 3 days of medication, the regimen is adjusted to 100μg qd. Treatment should continue until transfer out of the NICU or discharge, with a minimum duration of 7 days.
  Arms: Thyroid hormone replacement therapy
Drug: Euthyrox — Patient will not receive the oral levothyroxine sodium tablets.
  Arms: Non-thyroid hormone replacement therapy

SUMMARY:
Low levels of serum triiodothyronine (T3) thyroid hormones (T4) are a strong predictor of mortality and poor prognosis in critical care patients. Few reports, however, have focused on neurocritical patients.

Patients with severe neurological diseases often experience more complications and exhibit higher mortality rates, and many studies have provided evidence for a low T3/T4 state being an important prognostic indicator in such cases; Lieberman et al. found that 87% of individuals with severe traumatic brain injury have thyroid function below the mid-normal range. Other researchers showed that low T3 syndrome is a predictor of poor prognosis in cerebral infarction patients; their findings indicated the central hypothyroidism and disturbance of thyroid hormone metabolism were involved. Low T3 syndrome is common in patients with brain tumors and has been shown to be associated with shorter survival in glioma patients. Despite these observations, however, whether the thyroid hormone abnormalities in the critically ill are a physiological adaptation or a pathological change, and whether hormone replacement therapy (HRT) can benefit such patients, remain to be established.

As acute progression ceases, thyroid hormone levels may return to normal. This may imply that thyroid hormone supplements could improve the prognosis of patients with secondary hypothyroidism. Previous clinical studies have examined the effect of thyroid HRT on patients undergoing cardiac surgery; patients with malnutrition, heart failure, or acute renal failure; and premature infants with acute respiratory distress syndrome. Most of these past studies found no significant positive effects on prognosis, and no harmful effects either. Some smaller studies have demonstrated potential promise for the use of HRT; for example, one study showed that T3 supplementation in patients undergoing cardiac surgery could lead to less need for inotropic support and better hemodynamic parameters. There are no reports of thyroid HRT improving the prognosis of neurocritical patients with secondary hypothyroidism.

The application of hormone replacement therapy in the treatment of neurocritical patients with secondary hypothyroidism remains controversial.

This study aims to explore the safety and effectiveness of thyroid hormone replacement therapy in patients with spontaneous intracerebral hemorrhage and concomitant secondary hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

1. Admittance of neurocritical patients to the Neurological Intensive Care Unit (NICU) with a Glasgow Coma Scale (GCS) score of 3-8 and supratentorial hematoma volume >30 ml. The disease is limited to spontaneous intracerebral hemorrhage (supratentorial brain parenchyma, with or without hematoma rupture into the ventricle).
2. Age: 18-80 years old.
3. Onset within 24 hours.
4. Free T3 < 1.80 pg/ml or free T4 < 0.81 ng/dl within 7 days of onset, with or without TSH < 0.38 μIU/ml. (Specifically according to the critical values of different center laboratories' abnormal ranges).
5. Emergency head CT scan completed within 24 hours of onset.

Exclusion Criteria:

1. Organic thyroid lesions (subacute thyroiditis, chronic thyroiditis, post-thyroidectomy, thyroid radiation, hyperthyroidism), history of thyroid hormone oral replacement therapy within the past month.
2. Sella region lesions.
3. Baseline CT indicates irreversible brain herniation, expected survival period <30 days.
4. Severe systemic multiple injuries outside the nervous system.
5. Pregnant women.
6. Acute or chronic heart failure, arrhythmias, myocardial disease.
7. Only TSH levels decrease while free T3 and free T4 levels remain normal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
blood pressure | Day1、2、3、5、7（ 9:00 17:00 21:00）
  Systolic blood pressure in mmHg, diastolic blood pressure in mmHg, mean arterial pressure in mmHg, heart rate in beat per minute
cerebral blood flow dynamics | Day 7
  Cerebral blood volume in ml/100g; cerebral blood flow in ml/(100g·min)
Whether to use vasoactive vasopressors | Day 1 to 7
  Blood pressure in mmHg before and after using vasoactive vasopressors
neurological function | in 90 days
  modified Ranking Scale score (0 to 6 score, from better to worse)

SECONDARY OUTCOMES:
Days of the patients received intensive care | From date of randomization until the date of first documented progression or date of discharge from any cause, whichever came first, assessed up to 12 months
Mechanical ventilation time | From date of randomization until the date of first documented progression or date of discharge from any cause, whichever came first, assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China